CLINICAL TRIAL: NCT04221568
Title: The Comparison of Intrathecal Bupivacaine With Fentanyl and Levobupivacaine With Fentanyl for Labour Analgesia
Brief Title: Intrathecal Analgesia for Normal Labour
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Peter Elesha Roshdy, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Analgesia in normal labour
Record Dates: First submitted 2019-10-14; First posted 2020-01-09 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Labor Pain
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Intervention Model Description: multiparous parturients at term pregnancy (American society of anathesiologist physical status grade II)
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Bupivacaine-fentanyl — local anathetic&analgesic drugs
Drug: levobupivacaine-fentanyl — local anathetic&analgesic drugs

SUMMARY:
Primary outcome: Compare the duration of analgesia. Secondary outcome: analgesic potency of bupivacaine and fentanyl versus levobupivacaine and fentanyl.

DETAILED DESCRIPTION:
The pain of childbirth is the most severe pain any women can endure in their life time. Painful uterine contractions lead to maternal hyperventilation and increased catecholamine concentrations resulting im maternal and fetal hypoxemia.

Labour pain when unrelieved can have adverse effect on the course of labour as well as on the fetal wellbeing. An effective labour analgesia lead to better fetal and maternal outcome.

Although the gold standard in labour analgesia is utilization of epidural services which are widely used to provide pain-free labour in many parts of the world and and have the advantage of providing flexibility to meet the needs of each patient . Epidurals have long been associated with increased oxytocin use, increased fetal malposition, increased rates of instrumental and cesarian delivery, and longer labour .

The use of single-shot intrathecal low dose found to be effective . The advantages of this form of technique include the rapidity of onset and reliability, with minimal hemodynamic changes and motor block. Spinal block is cheaper as well as less technically challenging when compared to epidural and combined spinal epidural block. Intrathecal analgesia alone is useful when duration of labour can be reasonably estimated. Opioid combined with a small dose of local anesthetic provides rapid analgesia and dissipates when no longer needed.

Bupivacaine because of its least placental transfer, due to high protein binding and minimal motor block compared to sensory block in lower doses, has become the popular choice for labor analgesia. Addition of neuraxial lipid soluble opioids permitted reduction in the dose while maintaining effective analgesia and minimizing potential adverse effects on the progress of labor and lower extremity motor block .

Levobupivacaine is the S (-) enantiomer of racemic bupivacaine. Previous studies have shown that it exhibits a clinical profile similar to bupivacaine with the added advantage of less motor impairment .

ELIGIBILITY:
Inclusion Criteria:

1. singleton pregnancies
2. vertex presentation who will be in the active phase of labour with a cervical dilatation >4cm
3. normal fetal heart rate.

Exclusion Criteria:

* 1-Parturients with systemic diseases 2-Suspected cesarian section which include, in order of frequency, labor dystocia, abnormal or indeterminate (formerly, nonreassuring) fetal heart rate tracing, fetal malpresentation, multiple gestation, and suspected fetal macrosomia.
* 3 Fetus with known or suspected congenital abnormalities, and 4-Administration of parentral or oral analgesics before initiation of neuraxial analgesia will be excluded from the study.

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
Compare the duration of analgesia of bupivacaine and fentanyl versus levobupivacaine and fentanyl. | From2 to 8 hours. It is the time between the end of the spinal injection and the moment additional analgesia requested by parturients owing to the reappearance of labor pain was assessed by Visual Analog Scale for Pain (VAS Pain)
  Defined as the time between the end of the spinal injection and the moment additional analgesia requested by parturients owing to the reappearance of labor pain was assessed.

SECONDARY OUTCOMES:
Analgesic potency of bupivacaine and fentanyl versus levobupivacaine and fentanyl. | From2-8 hours. It is the time between the end of the spinal injection and the moment additional analgesia requested by parturients owing to the reappearance of labor pain was assessed by Visual Analog Scale for Pain (VAS Pain)
  Defined as the time between the end of the spinal injection and the moment additional analgesia requested by parturients owing to the reappearance of labor pain was assessed.

CONTACTS AND LOCATIONS:
Overall Officials: hamdy abbas, Study Director — Assiut University; wesam nashat, Study Director — Assiut University

REFERENCES:
- [Background] Brose D. [Pathology of the orofacial systems]. Zahntechnik (Berl). 1975 May;16(5):224-7. No abstract available. German. PMID 1077683